CLINICAL TRIAL: NCT00415220
Title: Comparison of Treatment Outcomes Between Chiropractic and Back Surgery for the Treatment of Sciatica Secondary to Lumbar Herniated Disc: A Prospective Randomized Controlled Trial.
Brief Title: Manipulation or Microdiscectomy For Sciatica? A Prospective Randomized Controlled Trial.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McMorland, Gordon, D.C. (Individual)
Collaborators: Foundation for Chiropractic Education and Research (FCER) (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FCER-99-10-04[99-03-03r]
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2006-12-22 (Estimated); Status verified 2006-12

CONDITIONS: Sciatica; Intervertebral Disk Displacement
Keywords: Chiropractic; Manipulation; Back surgery; Herniated lumbar disc; Sciatica; Lumbar microdiscectomy; Cost-effectiveness
MeSH Terms: conditions — Sciatica; Intervertebral Disc Displacement | interventions — Manipulation, Spinal

INTERVENTIONS:
Procedure: Spinal Manipulation, Microdiscectomy

SUMMARY:
The purpose of this study was to compare standardized chiropractic treatment (spinal manipulation) to back surgery (microdiscectomy) for patients with sciatica secondary to lumbar herniated disc refractory to medical management.

DETAILED DESCRIPTION:
Context: Operative management of lumbar radiculopathy caused by lumbar disc herniation (LDH) in patients refractory to medical management provides rapid and effective symptom relief. However, both short and long term benefits of surgery continue to be scrutinized.

Objective: To compare clinical efficacy of Chiropractic Treatment against Microdiscectomy in patients suffering from sciatica secondary to LDH.

Study Design: Prospective Randomized Controlled Clinical Trial allowing crossover, recruitment 2000-2004, 1 year follow-up.

Setting: Elective primary care physician referrals made directly to neurosurgical spine surgeons at the Foothills Hospital and Medical Centre, University of Calgary.

Patients: Forty consecutive consenting patients with sciatica from LDH refractory to at least three months of non-operative care and found appropriate for surgery.

Interventions: Surgical microdiscectomy or standardized chiropractic treatment. Crossover to the alternate treatment allowed after 3 months.

Main Outcome Measures: McGill Pain Score, Roland Morris Disability Index, Aberdeen Pain Scale, and SF-36 General Health Survey before treatment initiation and after 3, 6, 12, 24 and 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients presenting through elective referral by primary care physicians to one of the three participating spinal neurosurgeons (SC, SJD, RJH) between December 2000 and May 2004 were screened for symptoms of unilateral lumbar radiculopathy secondary to LDH at L3/4, L4/5 or L5/S1. Detailed surgical histories and physical examinations were performed on each referred patient by the consulting neurosurgeon and correlated with evidence of appropriate root compression on MR imaging. Patients who had failed at least 3 months of non-operative management including treatment with analgesics, lifestyle modification, physiotherapy, massage therapy and / or acupuncture, and who were felt appropriate for microdiscectomy by the neurosurgeon were asked to consider study participation.

Exclusion Criteria:

* Radicular symptoms < 3 months duration
* Major neurological deficits such as:

  * Cauda equina syndrome
  * Rapidly progressing neurological symptoms (e.g. foot drop)
* Substance abuse
* Hospitalization for intravenous or intramuscular narcotics
* Systemic or visceral disease (e.g. auto-immune diseases, major system failure)
* Hemorrhagic disorders, anticoagulation therapy
* Previous surgery at symptomatic level
* Concurrent chiropractic care at time of enrollment
* Prolonged use of systemic corticosteroids
* Osteopenia/Osteoporosis
* Spondylolisthesis grade III or IV
* Unable to read or speak English
* Age < 18
* Pregnancy
* Dementia or other cognitive impairment
* Unavailable for follow-up (geographic barriers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2000-01; Study Completion 2004-05

PRIMARY OUTCOMES:
McGill Pain Score
Roland Morris Disability Index
Aberdeen Pain Scale
SF-36 General Health Survey

CONTACTS AND LOCATIONS:
Overall Officials: Gordon McMorland, Principal Investigator
Locations (2):
- Canada (2):
  - National Spine Care, Calgary, Alberta
  - University of Calgary, Faculty of Medicine, Division of Neurosurgery, Calgary, Alberta